CLINICAL TRIAL: NCT06862882
Title: Impact of a Community-Based Primary Health Care Project on the Inappropriate Use of Emergency Medical System in Bergamo
Acronym: PHC-BG_EMS
Status: Recruiting | Type: Observational
Sponsor: Fondazione San Giuliano Onlus (Other)
Collaborators: FROM- Fondazione per la Ricerca Ospedale di Bergamo- ETS (FondazioneROM) (Unknown)
Responsible Party: Sponsor
Other Study IDs: PHC-BG_EMS study
Record Dates: First submitted 2025-02-25; First posted 2025-03-06 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Primary Health Care

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Behavioral: Community-Based Primary Health Care — Mediation between citizens and health workers to allow an orderly and appropriate use of social and health services

SUMMARY:
The goal of this study is to reduce the inappropriate use of the Emergency Medical System in Bergamo. The main question it aims to answer is: can a Community-Based Primary Health Care Project impact on the use of the Emergency Medical System in Bergamo? Monthly changes in urgent calls to the Emergency Medical System will be analysed.

ELIGIBILITY:
Inclusion Criteria:

* Urgent Emergency Medical System call

Exclusion Criteria:

* Non-urgent Emergency Medical System call

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Citizen who call Emergency Medical System
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of inappropriate access to Medical Emergency System | during the intervention
  Mediation between citizens and health workers to allow an orderly and appropriate use of social and health services and responding to the needs of the population, designing and implementing experimental activities to contrast the epidemic and promote health.

CONTACTS AND LOCATIONS:
Overall Officials: Mirco Nacoti, MD, Principal Investigator — Fondazione San Giuliano Onlus
Locations (1):
- Fondazione San Giuliano Onlus, Ciserano, Italy

IPD SHARING:
Plan to Share IPD: No